CLINICAL TRIAL: NCT05651776
Title: An Outpatient Physical Therapy and Golf Program Designed for Individuals With Movement Disorders
Brief Title: Golf, Physical Rehabilitation, and Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202202232
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease, Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Movement Disorders | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention of golf and rehab (Experimental): 2x/week x 6 weeks participation in a golf and PD rehab program
  Interventions: Other: Physical Therapy, Exercise

INTERVENTIONS:
Other: Physical Therapy, Exercise — Outpatient physical therapy intervention incorporating golf related assessment of skills and prescribed exercises including postural, balance, and club swing

SUMMARY:
The importance of physical activity for individuals with movement disorders, including Parkinson disease and Essential tremor, has been established. Barriers including patient engagement continue to limit effectiveness. Golf requires skills found challenging to individuals with movement disorders. This study seeks to assess the feasibility and effectiveness of an outpatient-based rehabilitation program incorporating golf skills and activities on functional measures and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of either PD, Parkinsonism, or ET. Subjects must also demonstrate functional deficits in at least one of the three categories (gait, transfers, balance) to be further assessed by the evaluating PT

Exclusion Criteria:

* Subjects will be excluded if they are unable to maintain standing balance with an assistive device, if they are non-ambulatory even with a device, if pain does not allow for subject participation, and if they are unable to follow instructions due to an underlying attentional or cognitive deficit.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Change in functional gait assessment | Scale completed at baseline and at 6 weeks of treatment
  Scale that measures ambulation quality

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Legacy, MD, Principal Investigator — UF Health Neurology
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No